CLINICAL TRIAL: NCT02083887
Title: A Phase I Study to Assess the Safety and Immunogenicity of ChAd63 ME-TRAP - MVA ME-TRAP Heterologous Prime-boost Vaccination Co-administered With EPI Vaccines in Gambian Infants
Acronym: VAC058
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Malaria Vectored Vaccines Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC058
Record Dates: First submitted 2014-02-28; First posted 2014-03-11 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Malaria
Keywords: Immune response; Vaccine; Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: ChAd63 ME-TRAP / MVA ME-TRAP at 16/24 weeks old (Active Comparator): ChAd63 ME-TRAP / MVA ME-TRAP. 15 infants aged 16 weeks at time of first vaccination vaccinated with ChAd63 ME-TRAP 5 x 10^10 vp (virus particles) intramuscular (IM) at 16 weeks and MVA ME-TRAP 1 x 10^8 pfu (plaque forming units) IM at 24 weeks.
  Interventions: Biological: ChAd63 ME-TRAP / MVA ME-TRAP
- Group 2: ChAd63 ME-TRAP / MVA ME-TRAP at 8/16 weeks old (Active Comparator): ChAd63 ME-TRAP / MVA ME-TRAP. 15 healthy infants aged 8 weeks at the time of first vaccination vaccinated with ChAd63 ME-TRAP 5 x 10^10 vp IM at 8 weeks and MVA ME-TRAP 1 x 10^8 pfu IM at 16 weeks
  Interventions: Biological: ChAd63 ME-TRAP / MVA ME-TRAP
- Group 3: ChAd63 ME-TRAP / MVA ME-TRAP at 1/8 weeks old (Active Comparator): ChAd63 ME-TRAP / MVA ME-TRAP. 15 healthy infants aged 1 week will be vaccinated with ChAd63 ME-TRAP 5 x 10^10 vp IM at 1 week and MVA ME-TRAP 1 x 10^8 pfu IM at 8 weeks.
  Interventions: Biological: ChAd63 ME-TRAP / MVA ME-TRAP
- Group 4: Control (No Intervention): 20 healthy infants aged 16, 8 and 1 weeks will be enrolled into this group. (Five infants will be randomised to each of Groups 1 and 2 respectively while 10 infants aged 1 week will be randomised to Group 3). All twenty infants will receive EPI vaccinations only.

INTERVENTIONS:
Biological: ChAd63 ME-TRAP / MVA ME-TRAP — Intramuscular administration of ChAd63 ME-TRAP 5 x 10^10 vp and MVA ME-TRAP 1 x 10^8 pfu
  Arms: Group 1: ChAd63 ME-TRAP / MVA ME-TRAP at 16/24 weeks old; Group 2: ChAd63 ME-TRAP / MVA ME-TRAP at 8/16 weeks old; Group 3: ChAd63 ME-TRAP / MVA ME-TRAP at 1/8 weeks old

SUMMARY:
Two vaccines, ChAd63 ME-TRAP and MVA ME-TRAP, are being tested to see if they will form a safe and effective vaccination strategy against malaria. The vaccines have been found to be well tolerated when tested in Gambian adults, young children and infants, who are at risk of severe malaria. Both vaccines will be given to participating infants at the same time as some EPI (Expanded Program on Immunization) vaccines, and assess whether they are safe and still helpful in making the body's defense system respond.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: 15 healthy infants aged 16 weeks at the time of enrolment with signed consent obtained from parents
* Group 2: 15 healthy infants aged 8 weeks at the time of enrolment with signed consent obtained from parents
* Group 3: 15 healthy infants aged 1 week at the time of enrolment with signed consent obtained from parents
* Group 4 (control): 20 healthy infants aged 16, 8 and 1 weeks at the time of enrolment with signed consent obtained from parents
* Groups 1 and 2: Receipt of all EPI vaccines according to schedule defined as follows: Bacillus Calmette-Guérin (BCG), and first dose of oral polio (OPV) and Hepatitis B vaccine within 2 weeks of birth; Penta, pneumococcal vaccine, OPV, rotavirus vaccine for Group 1 at 8 weeks +/- 2 weeks

Exclusion Criteria:

* Birth weight less than 2.5kg
* Significant antenatal, perinatal or early postnatal complications as judged by the PI or other delegated individual
* Any signs of acute illness as judged by the PI or other delegated individual
* Axillary temperature of greater than 37.5 °C
* Clinically significant congenital abnormalities as judged by the PI or other delegated individual
* Clinically significant history of skin disorder (psoriasis, contact dermatitis etc.), allergy, symptomatic immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness as judged by the PI or other delegated individual.
* Weight for age z-scores below 2 standard deviations of normal for age
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g. egg products, Kathon, neomycin, betapropiolactone.
* History of splenectomy
* Haemoglobin less than 10 g/dL at > 4 weeks of age or less than 13.0 g/dl at < 4 weeks of age.
* White cell count <5.0 x 109/L
* Serum Creatinine concentration greater than 60 micromol/L,
* Serum alanine aminotransferase (ALT) concentration greater than 45 U/L,
* Clinically significant jaundice
* Any other clinically significant laboratory abnormality as judged by the PI or other delegated individual
* Blood transfusion within one month of enrolment.
* History of vaccination with previous experimental malaria vaccines.
* Administration of any immunoglobulin less than two weeks before vaccination with the IMPs
* Current participation in another clinical trial, or within 12 weeks of this study.
* Any other finding which in the opinion of the PI or other delegated individual would increase the risk of an adverse outcome from participation in the trial.
* Likelihood of travel away from the study area
* Maternal HIV infection (a negative maternal HIV test will be required prior to study enrolment)
* Positive malaria antigen test at screening

Ages: 1 Week to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety of ChAd63 ME-TRAP / MVA ME-TRAP prime boost immunisation co-administered with EPI vaccines | Participants will be followed for the duration of the study, an expected average of 36 weeks
  Recording of all solicited and unsolicited local and systemic adverse events (including laboratory abnormalities considered adverse events) and the assessment of their causal relationships to the investigative medicinal products (IMPs).

SECONDARY OUTCOMES:
Immunogenicity of ChAd63 ME-TRAP / MVA ME-TRAP prime boost immunisation co-administered with EPI vaccines. | Participants will be followed for the duration of the study, an expected average of 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Afolabi, Principal Investigator — Medical Research Council Unit, The Gambia Unit
Locations (1):
- Medical Research Council Unit, Fajara, Banjul, The Gambia

REFERENCES:
- [Derived] Mensah VA, Roetynck S, Kanteh EK, Bowyer G, Ndaw A, Oko F, Bliss CM, Jagne YJ, Cortese R, Nicosia A, Roberts R, D'Alessio F, Leroy O, Faye B, Kampmann B, Cisse B, Bojang K, Gerry S, Viebig NK, Lawrie AM, Clarke E, Imoukhuede EB, Ewer KJ, Hill AVS, Afolabi MO. Safety and Immunogenicity of Malaria Vectored Vaccines Given with Routine Expanded Program on Immunization Vaccines in Gambian Infants and Neonates: A Randomized Controlled Trial. Front Immunol. 2017 Nov 20;8:1551. doi: 10.3389/fimmu.2017.01551. eCollection 2017. PMID 29213269